CLINICAL TRIAL: NCT01368757
Title: A Phase I/II Study of Lenalidomide in Patients With Chronic Myelomonocytic Leukemia
Brief Title: Lenalidomide in Patients With Chronic Myelomonocytic Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Prof. Dr. Richard Greil, Arbeitsgemeinschaft medikamentoese Tumortherapie
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_CMML 1; 2009-017147-33 (EudraCT Number)
Record Dates: First submitted 2011-05-09; First posted 2011-06-08 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Myelomonocytic Leukemia
Keywords: Chronic myelomonocytic leukemia; CMML; Lenalidomide; Revlimid
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Revlimid — Dose escalation 5mg - 10mg - 15mg - 20mg in cohorts of three patients
  The first step of phase I will be 5 mg lenalidomide in a daily regimen, the next step will be 10 mg in a daily regimen, the dosis of the following steps will be increased by 5 mg each until dose limiting toxicity (DLT) is reached.
  Phase II will be started at the MTD (1 dose step below DLT) and will be administered in a daily regimen.
  Other Names: lenalidomide; lenalidomid

SUMMARY:
In a phase I study the investigators plan to investigate safety and toxicity of lenalidomide in patients with Chronic Myelomonocytic Leukemia (CMML). A phase II study will be started once an optimal dose has been found. The primary endpoint will concern the efficacy of lenalidomide in patients with CMML according to the WHO diagnostic criteria.

ELIGIBILITY:
Inclusion Criteria:

1. CMML according to the WHO diagnostic criteria.
2. Understand and voluntarily sign an informed consent form.
3. Age >=18 years at the time of signing the informed consent form.
4. Able to adhere to the study visit schedule and other protocol requirements.
5. All previous cancer therapy must have been discontinued at least 4 weeks prior to treatment in this study. Patients carrying a somatic mutation involving the platelet derived growth factor receptor beta (PDGFRB) can be included if standard treatment with imatinib failed.
6. ECOG performance status of <= 2 at study entry.
7. Laboratory test results within these ranges:

   * Creatinine clearance > 30ml/min
   * AST (SGOT) and ALT (SGPT) <= 2.5 x ULN
8. Disease free of prior malignancies for >= 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
9. Female subjects of childbearing potential must:

   * Understand the study drug is expected to have a teratogenic risk
   * Agree to use two effective contraception
10. Male subjects must

    * Agree to use condoms
    * Agree not to donate semen
11. All subjects must

    * Agree to abstain from donating blood
    * Agree not to share study drug with another person

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other experimental drug or therapy within 28 days of baseline.
5. Known hypersensitivity to thalidomide.
6. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Any prior use of lenalidomide.
8. Concurrent use of other anti-cancer agents or treatments.
9. Known positive for HIV or infectious hepatitis, type A, B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-06; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 2 years
  This is a phase I/II, open-label, dose-escalation study of lenalidomide in patients with CMML. In phase I of the study the primary purpose is to determine the MTD. The purpose of phase II is to determine the response rate.

SECONDARY OUTCOMES:
Number and seriousness of adverse events to evaluate safety and tolerability | 4 years
  For both phases (phase I and II), secondary objectives are to evaluate safety, tolerability, efficacy and analysis of molecular markers.
Number of patients achieving transfusion independence | 4 years
  Phase II
Progression free survival, Overall survival | 4 years
  Phase II
Patients achieving cytogenetic response | 4 years
  Phase II; Cytogenetic response assessment requires 20 analyzable metaphases using conventional cytogenetic techniques, FISH may be used an a supplement to follow a specifically defined cytogenetic abnormality

CONTACTS AND LOCATIONS:
Overall Officials: Josef Thaler, MD, Study Director — Klinikum Wels-Grieskirchen GmbH; Sonja Burgstaller, MD, Study Director — Klinikum Wels-Grieskirchen GmbH
Locations (10):
- Austria (10):
  - Universitaetsklinik der PMU Salzburg, UK f. Innere Medizin III, Salzburg, Salzburg
  - Universitätsklinik f. Innere Medizin Graz, Klinische Abteilung f. Hämatologie, Graz, Styria
  - Universitätsklinik für Innere Medizin Innsbruck, Klinische Abteilung für Hämatologie und Onkologie, Innsbruck, Tyrol
  - Krankenhaus d. Barmherzigen Schwestern Linz, Interne I, Linz, Upper Austria
  - Krankenhaus der Elisabethinen Linz GmbH, 1. Interne, Linz, Upper Austria
  - AKH Linz, Innere Medizin 3, Zentrum für Hämatologie und medizinische Onkologie, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH, IV. Interne Abteilung, Wels, Upper Austria
  - MUW/ AKH Wien Univ. Klinik für Innere Medizin I, Abteilung für Hämatologie und Hämostaseologie, Vienna, Vienna
  - Hanusch Krankenhaus, 3. Med. Abtlg. Für Hämatologie und Onkologie, Vienna, Vienna
  - LKH Feldkirch, Interne E, Feldkirch, Vorarlberg